CLINICAL TRIAL: NCT02308631
Title: ENDOSCOPICALLY ASSISTED COLOSTOMY WITH COLOPEXY FOR CRITICALLY ILL PATIENTS WITHOUT GENERAL ANESTHESIA OR LAPAROTOMY. EXPERIMENTAL STUDY
Brief Title: Endoscopically Assisted Colostomy With Colopexy for Critically Ill Patients Without General Anesthesia or Laparotomy
Acronym: EACC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: LEONARDO ALFONSO BUSTAMANTE L (Unknown); MARIANNY NAZARETH SULBARAN N (Unknown); PAULO SAKAI (Unknown); EDUARDO MOURA (Unknown); CRISTIANO SAKAI (Unknown); CAIO SERGIO NAHAS (Unknown); CARLOS FREDERICO MARQUES (Unknown); IVAN CECONELLO (Unknown); SERGIO CARLOS NAHAS (Unknown)
Responsible Party: Principal Investigator, Leonardo Alfonso Bustamante, M.D. Colon and Rectal surgeon, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12267
Record Dates: First submitted 2014-09-24; First posted 2014-12-04 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-10

CONDITIONS: Colonic Neoplasms; Rectal Neoplasms; Fecal Incontinence
Keywords: Endoscopic, Colostomy, Colopexy
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colostomy with colopexy by endoscopy (Experimental): Colostomy with colopexy by endoscopy. 5 porks underwent endoscopic assisted colostomy with percutaneous colopexy. Animals were evaluated in post-operative days 1, 2, 5 and 7 Procedure/Surgery: ENDOSCOPICALLY ASSISTED COLOSTOMY WITH COLOPEXY
  Interventions: Procedure: ENDOSCOPICALLY ASSISTED COLOSTOMY WITH COLOPEXY

INTERVENTIONS:
Procedure: ENDOSCOPICALLY ASSISTED COLOSTOMY WITH COLOPEXY — The endoscope was manipulated until the light approached the pre-set for the use of transillumination site and puncture with the Loop Fixture II gastropexy kit

SUMMARY:
Indications for colostomy are rectal or anal cancer, diverticular disease, radiation enteritis, complex perirectal fistulas, anorectal trauma, severe incontinence, motility and functional disorders. It is frequently required in critically ill patients who may not be able to tolerate a laparotomy. Laparoscopic-assisted colostomy is an alternative method for colostomy without laparotomy, but require general anesthesia.

Additionally, percutaneous anterior colopexy under colonocopic control offers the possibility for improved and faster fixation of the anterior colonic wall to the anterior abdominal wall.

The objective of this study is to evaluate the feasibility of performing fecal diversion with the help of a colonoscope and colopexy, without the additional morbidity of abdominal exploration.

DETAILED DESCRIPTION:
The colonoscope will be passed transanally into the left colon. It will be identified the endoscopic transilluminating point to the abdominal wall. Percutaneous anterior colopexy will be performed, using a gastropexy device that is included in the percutaneous endoscopic gastrostomy (PEG) kit . This technique involves the placement of a threaded nylon fastener into the colon through a needle.

The endoscope will be manipulated until the light approaches the premarked site. A small skin disc will then be removed at this location and a loop colostomy will be made. The colonoscope will also be used as a guide to identify the proximal and distal limbs of the loop colostomy.

ELIGIBILITY:
Inclusion Criteria:

* good health and without surgery

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of the procedure | 7 days
  Feeding and mobilization of the animal, post procedure

SECONDARY OUTCOMES:
Number of animals with Adverse Events in the colostomy. | 7 days
  color of the edges and lost of function of the colostomy

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo A Bustamante, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Medicine School, Sao Paulo University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Mattingly M, Wasvary H, Sacksner J, Deshmukh G, Kadro O. Minimally invasive, endoscopically assisted colostomy can be performed without general anesthesia or laparotomy. Dis Colon Rectum. 2003 Feb;46(2):271-3. doi: 10.1007/s10350-004-6534-0. PMID 12576903
- [Result] Senapati A, Phillips RK. The trephine colostomy: a permanent left iliac fossa end colostomy without recourse to laparotomy. Ann R Coll Surg Engl. 1991 Sep;73(5):305-6. PMID 1929133
- [Result] Hellinger MD, Martinez SA, Parra-Davila E, Yeguez J, Sands LR. Gasless laparoscopic-assisted intestinal stoma creation through a single incision. Dis Colon Rectum. 1999 Sep;42(9):1228-31. doi: 10.1007/BF02238581. PMID 10496568